CLINICAL TRIAL: NCT02026349
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Efficacy and Safety of Favipiravir in Adult Subjects With Uncomplicated Influenza (T705US316)
Brief Title: Phase 3 Efficacy and Safety Study of Favipiravir for Treatment of Uncomplicated Influenza in Adults - T705US316
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MDVI, LLC (Industry)
Collaborators: MediVector, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T705US316; 2013-002149-13 (EudraCT Number)
Record Dates: First submitted 2013-12-19; First posted 2014-01-03 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: influenza; flu; fever; cough; body aches; headache; nasal congestion; body pains; sore throat; fatigue; T-705; favipiravir; favor; flu symptoms
MeSH Terms: conditions — Influenza, Human; Fever; Cough; Headache; Nasal Obstruction; Pharyngitis; Fatigue | interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- favipiravir (Active Comparator)
  Interventions: Drug: favipiravir
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: favipiravir — Administered twice daily over 5 consecutive days for a total of 10 doses.
  * Day 1: 1800 mg twice daily (loading doses)
  * Days 2 through 5: 800 mg twice daily
  Other Names: T-705
  Arms: favipiravir
Drug: Placebo — Administered twice daily over 5 consecutive days for a total of 10 doses.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if favipiravir is effective in reducing the time to resolution of influenza symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to determine if a 5-day regimen of favipiravir reduces the time to alleviation of influenza symptoms, resolution of fever, and viral shedding, in subjects with uncomplicated influenza compared to no treatment (e.g. placebo).

ELIGIBILITY:
Inclusion Criteria:

* At time of enrollment has 2 or more of the following symptoms (moderate to severe in intensity) that began 48 hours or less prior to the anticipated start of dosing with study medication: cough, sore throat, headache, nasal congestion, body aches and pains, fatigue
* Has a fever at the first visit or in the 6 hours prior if antipyretics were taken, defined as: ≥ 38.0°C (≥ 100.4°F) if < 65 years old; or ≥ 37.8°C (≥ 100.0°F) if ≥ 65 years old
* Tests positive for influenza A or B during the 48 hours between onset of symptoms and anticipated dosing with study medication as confirmed by RAT or PCR testing (study or non-study procedure); or per Investigator and Medical Monitor discretion in the event there is a known influenza outbreak circulating in the community or the subject has been in close contact with a person who was recently confirmed to have laboratory-confirmed influenza
* Willing to adhere to strict contraceptive measures throughout study and for 3 months following last dose of study medication

Exclusion Criteria:

* Female subjects who are pregnant, currently breast-feeding, or have a positive pregnancy test at Screening
* Has taken an anti-influenza drug, or received any live attenuated influenza vaccine within 4 weeks prior to signing the informed consent
* Has underlying chronic respiratory disease; includes bronchial asthma if currently experience asthma symptoms, requires current asthma treatment, or has had an asthma attack in the past year
* Is suspected of having bacterial respiratory infection (i.e., expectoration of purulent or mucopurulent sputum and/or infiltrate in lung observed on chest x ray, or is on antibiotics for pulmonary disease) at start of study
* Has a history of gout or is under treatment for: gout or hyperuricemia; hereditary xanthinuria; hypouricemia or xanthine calculi of the urinary tract
* Has a history of hypersensitivity to an anti-viral nucleoside-analog drug targeting a viral RNA polymerase
* Current use of adrenocorticosteroids (except topical preparation) or immunosuppressive drugs
* Has an allergy or contraindication to use of acetaminophen (paracetamol)
* Has a serious chronic disease, history of alcohol or drug abuse within preceding 2 years, psychiatric illness not well controlled (not on stable regimen > 1 year), or is deemed by the Investigator to be ineligible for any reason
* Previously participated in a clinical trial of favipiravir (T-705)
* Has renal insufficiency requiring hemodialysis or continuous ambulatory peritoneal dialysis (CAPD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time to alleviation of all primary influenza symptoms and fever | 21 days
  Time from the start of study treatment until alleviation of all primary influenza symptoms (i.e. cough, sore throat, headache, nasal congestion, body aches and pains, fatigue) and to resolution of fever. Subjects will be considered to have symptoms alleviated if individual symptoms are no greater than mild and are confirmed to be no greater than mild at least 21.5 hours later. Similarly, resolution of fever is defined as temperature (oral) measurements to be < 38.0°C (<100.4°F) for subjects < 65 years old and < 37.8°C (100.0°F) for subjects ≥ 65 years old, and measurements are confirmed at least 21.5 hours later. For the primary endpoint, the time periods of alleviation/fever resolution must be concurrent for symptoms and temperature.

SECONDARY OUTCOMES:
Time to alleviation each of the primary influenza symptoms and fever | 21 days
  Time from the start of study treatment until alleviation of each of the following influenza symptoms (cough, sore throat, headache, nasal congestion, body aches and pains, and fatigue) and to resolution of fever. Subjects will be considered to have symptoms alleviated if individual symptoms are no greater than mild and are confirmed to be no greater than mild at least 21.5 hours later. Similarly, resolution of fever is defined as temperature (oral) measurements to be < 38.0°C (<100.4°F) for subjects < 65 years old and < 37.8°C (100.0°F) for subjects ≥ 65 years old, and measurements are confirmed at least 21.5 hours later. Additional analyses of symptoms, including assessment of the impact of relevant covariates, will be specified in the Statistical Analysis Plan.
To characterize the PK of favipiravir when used under clinical conditions | 21 days
  Population PK analysis of favipiravir with assessment of maximum plasma concentration (Cmax), minimum plasma concentration (Cmin), and total daily exposure AUC(0-24h) on Visits 1, 2, 3, 4 and 5

OTHER OUTCOMES:
Changes in viral load | 15 days
  Changes in viral load (nasopharyngeal swabs) as measured by quantitative polymerase chain reaction (qPCR) and in the determination of median tissue culture infective dose (TCID50), from nasopharyngeal swabs at Visits 2, 3, 4, and 5; and log-transformed viral load (by qPCR and TCID50) area under the curves (AUCs).
Safety | 21 days
  Adverse events and clinical laboratory tests for systemic safety including hematology, clinical chemistry, and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Carol Epstein, MD, Study Director — MediVector, Inc.
Locations (188):
- United States (51):
  - Birmingham, Alabama
  - Hunstville, Alabama
  - Hot Springs, Arkansas
  - Los Angeles, California
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Tustin, California
  - Upland, California
  - Colorado Springs, Colorado
  - Hamden, Connecticut
  - Bradenton, Florida
  - Brooksville, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Lakeland Hills, Florida
  - Miami, Florida
  - Saint Cloud, Florida
  - South Miami, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Snellville, Georgia
  - Bardstown, Kentucky
  - Monroe, Louisiana
  - Opelousas, Louisiana
  - Flint, Michigan
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Hickory, North Carolina
  - Morganton, North Carolina
  - Winston-Salem, North Carolina
  - Lansdale, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Smithfield, Pennsylvania
  - Uniontown, Pennsylvania
  - Gaffney, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Simpsonville, South Carolina
  - Arlington, Texas
  - Austin, Texas
  - Carrollton, Texas
  - Forth Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Arlington, Virginia
  - La Crosse, Wisconsin
- Bedford Park, South Australia, Australia
- Belgium (10):
  - Deurne, Antwerpen
  - Brussels, Brussels Capital
  - Gozée, Hainaut
  - Mont-sur-Marchienne, Hainaut
  - Halen, Limburg
  - Ham, Limburg
  - Chenée, Liège
  - Deurne
  - Gribomont
  - Linkebeek
- Bulgaria (18):
  - Gabrovo, Gabrovo
  - Haskovo, Haskovo
  - Plovdiv, Plovdiv
  - Smolyan, Smolyan
  - Sofia, Sofia-Grad
  - Varna, Varna
  - Veliko Tarnovo, Veliko Tarnovo
  - Burgas
  - Gabrovo
  - Plovdiv
  - Rousse
  - Samokov
  - Sevlievo
  - Sliven
  - Smolyan
  - Sofia
  - Varna
  - Veliko Tarnovo
- Hungary (8):
  - Balassagyarmat
  - Budapest
  - Csongrád
  - Debrecen
  - Gödöllő
  - Gyula
  - Nyíregyháza
  - Zalaegerszeg
- Netherlands (7):
  - Nijverdal, Overijssel
  - Hoogvliet, South Holland
  - Lieshout
  - Nijverdal
  - Rotterdam
  - The Hague
  - Zwijndrecht
- New Zealand (4):
  - Auckland, North Island
  - Christchurch, South Island
  - Hamilton, Waikato Region
  - Tauranga
- Poland (16):
  - Torun, Kuyavian-Pomeranian Voivodeship
  - Tarnów, Lesser Poland Voivodeship
  - Oleśnica, Lower Silesian Voivodeship
  - Wroclaw, Lower Silesian Voivodeship
  - Świdnik, Lublin Voivodeship
  - Lodz, Lódzkie
  - Zgierz, Lódzkie
  - Łosice, Masovian Voivodeship
  - Dębica, Podkarpackie Voivodeship
  - Rzeszów, Podkarpackie Voivodeship
  - Katowice, Silesian Voivodeship
  - Katowice
  - Krakow
  - Lódz
  - Ostróda
  - Oświęcim
- Russia (10):
  - Arkangelsk
  - Kazan'
  - Moscow
  - Novosibirsk
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Tomsk
  - Vladimir
  - Yaroslavl
- South Africa (22):
  - Bloemfontein, Free State
  - Bryanston, Gauteng
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Sophiatown, Johannesburg, Gauteng
  - Soweto, Gauteng
  - Dundee, KwaZulu-Natal
  - eManzimtoti, KwaZulu-Natal
  - Middelburg, Mpumalanga
  - Witbank, Mpumalanga
  - Cape Town, Western Cape
  - Paarl, Western Cape
  - Worcester, Western Cape
  - Cape Town
  - Durban
  - eMkhomazi
  - Johannesburg
  - Krugersdorp
  - Potchefstroom
  - Pretoria
  - Sophiatown, Johannesburg
  - Welkom
- Spain (10):
  - Alicante, Alicante
  - Benidorm, Alicante
  - Orihuela, Alicante
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Castellon, Castellón
  - Barcelona, Catalonia
  - Llançà, Girona
  - Tarragona, Tarragona
  - Barcelona
- Sweden (8):
  - Malmo, Skåne County
  - Stockholm, Södermanland County
  - Uppsala, Uppsala Ian
  - Gothenburg, Västra Götaland County
  - Karlskrona
  - Linköping
  - Malmo
  - Uppsala
- Turkey (Türkiye) (10):
  - Diyarbakır, Diyarbakır
  - Izmir, İzmir
  - Konya, Konya
  - Trabzon, Trabzon
  - Ankara
  - Düzce
  - Erzurum
  - Eskişehir
  - Izmir
  - Samsun
- Ukraine (13):
  - Chernivtsi, Chernivtsi Oblast
  - Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kharkiv, Kharkivs’ka Oblast’
  - Kyiv, Kyïvs'ka Oblast
  - Kyiv, Kyïv
  - Odesa, Odesa Oblast
  - Ternopil, Ternopil Oblast
  - Vinnytsia, Vinnytsia Oblast
  - Kharkiv
  - Kherson
  - Kyiv
  - Poltava
  - Sumy

REFERENCES:
- [Derived] Hayden FG, Lenk RP, Stonis L, Oldham-Creamer C, Kang LL, Epstein C. Favipiravir Treatment of Uncomplicated Influenza in Adults: Results of Two Phase 3, Randomized, Double-Blind, Placebo-Controlled Trials. J Infect Dis. 2022 Nov 11;226(10):1790-1799. doi: 10.1093/infdis/jiac135. PMID 35639525